CLINICAL TRIAL: NCT01950182
Title: A Multicentre, Randomized Study of Trastuzumab Combined With Chemotherapy or Endocrine Therapy as the First Line Treatment for Patients With Metastatic Luminal B2 Breast Cancer Subtype
Brief Title: Trastuzumab Combined With Chemotherapy or Endocrine Therapy to Treat Metastatic Luminal B2 Breast Cancer
Acronym: SYSUCC-002
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, unYat-senU, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-002
Record Dates: First submitted 2013-09-18; First posted 2013-09-25 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: Luminal B2 subtype; First line treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Tamoxifen; Aromatase Inhibitors; Capecitabine; Vinorelbine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palliative chemotherapy (Active Comparator): Chemotherapy combined with trastuzumab. Chemotherapy could use the following drugs such as capecitabine , Vinorelbine, or Gemcitabine.
  Interventions: Drug: Chemotherapy combined with trastuzumab
- Palliative endocrine therapy (Experimental): Endocrine therapy combined with trastuzumab. Endocrine therapy could use tamoxifen or aromatase inhibitors including anastrozole, letrozole, or exemestane.
  Interventions: Drug: Endocrine therapy combined with trastuzumab

INTERVENTIONS:
Drug: Endocrine therapy combined with trastuzumab — Tamoxifen or aromatase inhibitors (Anastrozole, Letrozole, or Exemestane) combined with trastuzumab
  Other Names: Tamoxifen; aromatase inhibitors; trastuzumab
  Arms: Palliative endocrine therapy
Drug: Chemotherapy combined with trastuzumab — Capecitabine , Vinorelbine, or Gemcitabine combined with trastuzumab
  Other Names: Capecitabine; Vinorelbine; Gemcitabine; trastuzumab
  Arms: Palliative chemotherapy

SUMMARY:
The primary objective of this study is to compare progression-free survival (PFS) of patients with metastatic Luminal B2 breast cancer subtype randomised to treatment with Trastuzumab Combined With Chemotherapy or Endocrine Therapy.

DETAILED DESCRIPTION:
This is a non-inferiority study to examine Trastuzumab combined with chemotherapy or endocrine therapy in patients with metastatic Luminal B2 breast cancer subtype. The main purposes of this study are to test the safety and clinical benefit of Trastuzumab combined with chemotherapy or endocrine therapy in treating Luminal B2 breast cancer (hormone receptor positive and human epidermal growth factor receptor (HER2) positive or amplification). This multicentre, randomized study is designed to recruit up to 392 subjects to identify 196 research subjects for each study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Patients with an Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.
3. Histologically confirmed metastatic or local recurrence of breast cancer.
4. ER positive and/or progesterone receptor (PR) positive, HER-2+ defined as immuno-histochemistry3+ staining or FISH+.
5. Prior adjuvant Trastuzumab therapy is permitted, but disease-free interval (DFI) must be more than 12 months.
6. Patients must have measurable or evaluable disease.
7. Adequate bone marrow reserve with neutrophils > 1000 and platelets > 100,000.
8. Adequate renal function with serum creatinine < 2.0.
9. Adequate hepatic reserve with serum bilirubin < 2.0, alanine transaminase(ALT) < 3 times the upper limit of normal, and alkaline phosphatase < 5 times the upper limit of normal.
10. Adequate cardiac reserve with at least 45% of Left ventricular ejection fraction (LVEF) by echocardiogram.
11. Able to give informed consent.
12. Life expectancy of at least 12 weeks.

Exclusion Criteria:

1. Pregnant or breast feeding.
2. ECOG score ≧2
3. DFI <12 months.
4. LVEF < 45% by echocardiogram.
5. Uncontrolled medical problems.
6. Evidence of active acute or chronic infection.
7. Hepatic, renal, or bone marrow dysfunction as detailed above.
8. Concurrent malignancy or history of other malignancy within the last five years except as noted above.
9. Known severe hypersensitivity to Trastuzumab.
10. Patients were unable or unwilling to comply with program requirements.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2013-09-16 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 36 months
  The interim analysis and the final analysis are expected ot occur 18 and 36 months after the end of recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-yu Yuan, MD, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No